CLINICAL TRIAL: NCT03670966
Title: A Phase I/II Study Evaluating Escalating Doses of 211At-Labeled Anti-CD45 MAb BC8-B10 (211At-BC8-B10) Followed by Related Haplo-Identical Allogeneic Hematopoietic Cell Transplantation for High-Risk Acute Leukemia or Myelodysplastic Syndrome (MDS)
Brief Title: 211At-BC8-B10 Followed by Donor Stem Cell Transplant in Treating Patients With Relapsed or Refractory High-Risk Acute Leukemia or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1003349; 10060 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); NCI-2018-01788 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA078902 (NIH)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia in Remission; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome With Excess Blasts; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Refractory Mixed Phenotype Acute Leukemia; Hematopoietic and Lymphoid Cell Neoplasm
Keywords: Lymphoid Leukemia; Myeloid and Monocytic Leukemia; Other Hematopoietic
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Hematologic Neoplasms; Leukemia, Lymphoid; Leukemia, Monocytic, Acute | interventions — Cyclophosphamide; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation; Mycophenolic Acid; pegylated granulocyte colony-stimulating factor; fludarabine phosphate; Tacrolimus; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (211At-BC8-B10, chemotherapy, TBI, MMF, G-CSF) (Experimental): PREPARATIVE REGIMEN: Patients receive astatine At 211 anti-CD45 monoclonal antibody BC8-B10 infusion over 6-8 hours on day -8, fludarabine IV over 30 minutes on days -6 to -2, and cyclophosphamide IV over 1 hour on days -6 and -5. Patients also undergo TBI on day -1.
  TRANSPLANT: Patients undergo PBSC or bone marrow transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID on days 5-35, and tacrolimus IV over 1-2 hours (changed to PO once tolerated) on days 5-180 with taper beginning on day 84 per physician discretion. Patients also begin G-CSF IV or SC on day 5 to continue until ANC > 1000/mm^3 x 3 days.
  Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Biological: Astatine At 211 Anti-CD45 Monoclonal Antibody BC8-B10; Drug: Cyclophosphamide; Radiation: Total-Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Bone Marrow Transplantation; Drug: Mycophenolate Mofetil; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Drug: Fludarabine Phosphate; Drug: Tacrolimus; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Astatine At 211 Anti-CD45 Monoclonal Antibody BC8-B10 — Given via infusion
  Other Names: At 211 MAb BC8-B10; APAMISTAMAB-B10-ASTATINE AT-211
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; Asta B 518; B-518; WR-138719
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; SCT_TBI; Whole Body Irradiation; Whole-Body Irradiation; TBI
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC transplantation
  Other Names: PBPC transplantation
Procedure: Bone Marrow Transplantation — Undergo bone marrow transplant
  Other Names: Bone Marrow Grafting; BMT
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: 115007-34-6; MMF; Cellcept
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given IV or SC
  Other Names: 143011-72-7; Recombinant Colony-Stimulating Factor 3; rhG-CSF
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara; Fludarabine-5''-Monophosphate; SH T 586
Drug: Tacrolimus — Given IV or PO
  Other Names: Prograf; Protopic; FK 506; FK-506; Tacforius
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow biopsy and aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase I/II trial studies the side effects and best dose of a radioactive agent linked to an antibody (211At-BC8-B10) followed by donor stem cell transplant in treating patients with high-risk acute leukemia or myelodysplastic syndrome that has come back (recurrent) or isn't responding to treatment (refractory). 211At-BC8-B10 is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving chemotherapy and total body irradiation before a stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can attack the body's normal cells, called graft versus host disease. Giving cyclophosphamide, mycophenolate mofetil, and tacrolimus after a transplant may stop this from happening.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of astatine At 211 anti-CD45 monoclonal antibody BC8-B10.

PREPARATIVE REGIMEN: Patients receive astatine At 211 anti-CD45 monoclonal antibody BC8-B10 infusion over 6-8 hours on day -8, fludarabine intravenously (IV) over 30 minutes on days -6 to -2, and cyclophosphamide IV over 1 hour on days -6 and -5. Patients also undergo TBI on day -1.

TRANSPLANT: Patients undergo peripheral blood stem cell (PBSC) or bone marrow transplant on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO three times daily (TID) on days 5-35, and tacrolimus IV over 1-2 hours (changed to PO once tolerated) on days 5-180 with taper beginning on day 84 per physician discretion. Patients also begin granulocyte colony-stimulating factor (G-CSF) IV or subcutaneously (SC) on day 5 to continue until absolute neutrophil count (ANC) > 1000/mm^3 x 3 days.

Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at day 100, and at 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have AML, ALL, high-risk MDS, or MPAL (also known as biphenotypic) meeting one of the following descriptions:

  * AML, ALL, or MPAL in first remission with evidence of measurable residual disease (MRD) by flow cytometry;
  * AML, ALL, or MPAL beyond first remission (i.e., having relapsed at least one time after achieving remission in response to a treatment regimen);
  * AML, ALL, or MPAL representing primary refractory disease (i.e., having failed to achieve remission at any time following one or more prior treatment regimens);
  * AML evolved from myelodysplastic or myeloproliferative syndromes;
  * MDS expressed as refractory anemia with excess blasts (RAEB)
  * Chronic myelomonocytic leukemia (CMML) by French-American-British (FAB) criteria.
* Patients not in remission must have CD45-expressing leukemic blasts. Patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative (because in remission patients, virtually all antibody binding is to non-malignant cells which make up >= 95% of nucleated cells in the marrow).
* Patients must be >= 18 and =< 75 years of age.
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed).
* Patients must have an estimated creatinine clearance greater than 50/ml per minute by the following formula (Cockcroft-Gault). Serum creatinine value must be within 28 days prior to registration.
* Bilirubin < 2 times the upper limit of normal.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times the upper limit of normal.
* Eastern Cooperative Oncology Group (ECOG) < 2 or Karnofsky >= 70.
* Patients must be free of uncontrolled infection.
* Patients with prior non-myeloablative or reduced-intensity conditioning allogeneic-HCT must have no evidence of ongoing GVHD and be off all immunosuppression for at least 6 weeks at time of enrollment.
* Patients must have normal elastography.
* If ferritin is elevated, patient must have less than 7 mg/g liver iron concentration on liver T2 magnetic resonance imaging (MRI).
* Patients should have an official gastrointestinal (GI) consult prior to the transplant for full evaluation.
* Patients must have a related donor who is identical for one HLA haplotype and mismatched at the HLA-A, -B or DRB1 loci of the unshared haplotype with the exception of single HLA-A, -B or DRB1 mismatches.
* DONOR: Donors must meet HLA matching criteria as well as standard Seattle Cancer Care Alliance (SCCA) criteria for PBSC or bone marrow donation. Preference should be given to donors who are mismatched at the HLA-A, -B and -DRB1 loci.

Exclusion Criteria:

* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects.
* Left ventricular ejection fraction < 45%.
* Corrected diffusion capacity of the lung for carbon monoxide (DLCO) < 35% or receiving supplemental continuous oxygen. When pulmonary function tests (PFTs) cannot be obtained, the 6-minute walk test (6MWT, also known as exercise oximetry) will be used: Any patient with oxygen saturation on room air of < 89% during a 6MWT will be excluded
* Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease.
* Patients who are known to be seropositive for human immunodeficiency virus (HIV).
* Perceived inability to tolerate diagnostic or therapeutic procedures.
* Active central nervous system (CNS) leukemia at time of treatment.
* Patients with prior myeloablative allogeneic-HCT.
* Women of childbearing potential who are pregnant (beta human chorionic gonadotropin [B-HCG]+) or breast feeding.
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant.
* Inability to understand or give an informed consent.
* Allergy to murine-based monoclonal antibodies.
* Known contraindications to radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Toxicity: Proportion of patients who develop grades III/IV Bearman regimen-related toxicity | Up 100 days after hematopoietic cell transplantation (HCT)
  Proportion of patients who develop grades III/IV Bearman regimen-related toxicity.

SECONDARY OUTCOMES:
Achievement of remission | Up to 2 years
Rate of engraftment | Up to 2 years
Donor chimerism | At days 28, 56, 84, 180, and at 1 year
Non-relapse mortality (NRM) | Up to 2 years
Number of patients experiencing Immune reconstitution | Up to 2 years
Number of patients experiencing Number of Grade II-IV acute graft versus host disease (GVHD) | Up to 2 years
Number of patients experiencing Moderate/severe chronic GVHD | Up to 2 years
Overall survival | Up to 100 days
Disease-free survival | Up to day 100

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Vo, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No